CLINICAL TRIAL: NCT04150718
Title: Investigating the Role of Slow-wave Activity as a Marker of Impaired Plasticity in Major Depressive Disorder
Brief Title: Role of Slow-wave Activity and Plasticity in MDD
Acronym: SWIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 832986; K23MH118580 (NIH)
Record Dates: First submitted 2019-10-07; First posted 2019-11-05 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with Major Depressive Disorder (Experimental): Subjects who get assigned to this group will undergo a Diagnostic and Statistical Manual for Mental Disorders (SCID) assessment to determine is they meet criteria for MDD.
  Interventions: Behavioral: slow-wave disruption
- Control (Active Comparator): Subjects who get assigned to this group will undergo a Diagnostic and Statistical Manual for Mental Disorders (SCID) assessment to determine they do not meet criteria for MDD.
  Interventions: Behavioral: slow-wave disruption

INTERVENTIONS:
Behavioral: slow-wave disruption — A tone will be played through a speaker mounted over the bed that disrupts subjects while they are in slow-wave sleep. The tone will not be loud enough to wake up.

SUMMARY:
The hypothesis underlying this proposal is that deficits of synaptic plasticity underlie the slow-wave activity (SWA) abnormalities observed n major depressive disorder (MDD), and that manipulating SWA may serve to circumvent these deficits by facilitating an increase in synaptic strength via the inhibition of synaptic down-scaling, thereby improving plasticity and mood.

DETAILED DESCRIPTION:
VISIT 1: Screening. Participants who meet initial inclusion criteria via phone screen will be invited to the laboratory for an in-person screening visit that includes additional screening (e.g. Medical history, TMS eligibility, hearing test for SW disruption procedure), and a structured clinical interview to determine final study eligibility. All subjects will receive verbal and written explanation of the general goals and risks of the study and will sign an informed consent. At this session, participants will also have the opportunity to become acquainted with the TMS and SW disruption procedures. In the case that remote visits are being utilized, such as during the COVID-19 pandemic, this will be separated into a virtual visit (consent, clinical interview, etc. - anything that can be conducted remotely will be) and an in-person visit (hearing test, TMS demonstration). Participants will also choose two dates, at least two nights apart and at most separated by two weeks, for the in-lab visits.

At-home Sleep Recording. For 7 days prior to the in-lab study visits, participants will be asked to keep a consistent at-home sleep schedule, based on habitual rise time (e.g., 10:30 PM - 6 AM). Participants will also consent to refraining from napping, using alcohol and drugs, and limiting caffeine use to one caffeinated beverage before noon throughout the study. These procedures will be confirmed using actigraphy, and sleep diary. Actigraphy provides a validated measure of sleep-wake patterns based on light and activity levels utilizing a wrist-watch like device (Actiwatch 2 and Actiwatch Spectrum Pro, Philips Respironics, Inc.). Sleep diaries will be used to document bedtime and rise time, and several other sleep parameters. Participants will also be asked to note if actigraphs were removed, for how long and for what purpose. Sleep diaries will be completed via the REDCap web-based application if participants have consistent Internet access. Paper and pencil versions of sleep diaries will also be available. Study staff will compare across these methods to verify adherence to study guidelines prior to the in-lab study.

VISIT 2: Baseline Night. Visit 2 and Visit 3 occur on two separate days, in a counterbalanced design to ensure no order or learning effects. The following procedure description will occur in half of participants where Visit 2 precedes Visit 3; however identical procedures will be used for the remaining half of participants where Visit 3 will precede Visit 2. Participants will arrive at the Clinical Research Center for Sleep (CRCS) at 8pm on Visit 2. Following their arrival and orientation, EEG electrodes will be applied. Participants sleep will then be monitored overnight. In the morning, participants will have their blood drawn, and after a light breakfast, the HAM-D will be administered, and then participants will be asked to fill out mood questionnaires (BDI, VAS, PANAS, KSS), and complete a battery of tasks including memory tasks, and resting EEG. They will then be accompanied to the Richards Building to complete the TMS protocol, before returning to the CRCS.

VISIT 3: Slow-wave Disruption. Procedures for Visit 3 are identical for those for Visit 2, with the exception of the following: Utilizing real-time EEG monitoring during sleep, left (C3) and right central (C4) channels will be continuously inspected. Whenever two delta waves (14 Hz; 75 V) appear within 15 seconds, an acoustic stimulus (i.e. tone; frequency = 1000 Hz; intensity = 20100 dB) will be administered through a speaker mounted above the bed, beginning with the lowest intensity (20 dB) and increased by 5 dB intervals if no response occurs (sleep stage shift, K complex, EEG desynchronization, mixed and fast frequency, alpha burst, muscle tone increase, slow eye movements). Utilizing this methodology, the type and incidence of tones played will be tailored to each participant to suppress slow waves without arousing the subject. Disruption of SWA will take place without waking the subject or decreasing total sleep time. The selective SW disruption procedure has been described in detail elsewhere.

TMS The TMS system is housed in the Richards Biomedical Building. Only individuals trained by the IDE sponsor (Desmond Oathes, Ph.D.) and Center Director (Yvette Sheline, M.D.) will dispense TMS. Since all TMS procedures are being conducted in Dr. Sheline's lab, all plans for receipt, storage, labelling, dispensing, returning of failed devices, and destruction will fall under the center's SOPs.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-50
* Right handed
* English speaking
* Normal cognition
* Normal or corrected-to-normal vision and hearing
* Current depression as assessed on the SCID and Hamilton Rating Scale for Depression
* Stable, normally-time sleep-wake cycles as determined by interview, 1-week daily sleep log and 1-week wrist actigraphy evidence

Exclusion Criteria:

* Current or prior medical condition
* History of stroke, epilepsy, brain aneurysm clip or head injury causing unconsciousness
* Implanted devices (i.e. aneurysm clip or cardiac pacemaker)
* Sleep disorders other than insomnia
* History of bipolar disorder, delirium, dementia, amnestic disorder, schizophrenia and other psychotic disorders
* No history of depression for the control group.
* For women, pregnancy will exclude participation.
* Lifetime history of electroconvulsive therapy
* travel beyond 2 time zones in the 2 months before study
* Unwillingness to refrain from using alcohol or caffeine during the study

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldschmied, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Department of Psychiatry, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
All subject data will be de-identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- Unassigned Due to Ineligibility/Withdrawal: These individuals were either deemed ineligible or withdrew prior to the diagnostic interview and were therefore unassigned to a diagnostic group
Period: Overall Study
Arm/Group | Control | Subjects With Major Depressive Disorder | Unassigned Due to Ineligibility/Withdrawal
Started | 24 | 42 | 11
Completed | 20 | 33 | 0
Not Completed | 4 | 9 | 11
Not completed — Withdrawal by Subject | 2 | 7 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Ineligible | 1 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Ineligible/Withdrew: Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results.
- Total: Total of all reporting groups
Arm/Group | Subjects With Major Depressive Disorder | Control | Ineligible/Withdrew | Total
Number analyzed (Participants) | 33 | 20 | 11 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 20 | 11 | 64
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (5.32) | 32.68 (7.03) | NA (NA) — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | 31.63 (6.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | NA — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 13 | 10 | NA — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | NA — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | 1 | 4 | NA — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | 0 | 0 | NA — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | 5 | 3 | NA — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | 26 | 13 | NA — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | 1 | 0 | NA — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | NA — Results are reported per Arm/Group, but data from participants who were ineligible or withdrew were not included in the analysis, as we were not able to collect data from these participants. Therefore, these Arms/Groups are not represented in the reported results. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 33 | 20 | 11 | 53

OUTCOME MEASURES:

1. Primary Outcome: Compare Indices of Net Synaptic Strength (Transcranial Magnetic Stimulation Evoked Potentials) in Individuals With MDD to Healthy Controls
Description: Transcranial magnetic stimulation evoked potentials (MEP) - Measure of the amplitude of muscle movement from hand following TMS
Time Frame: one month
Population: Due to technical problems with the TMS protocol, data from N=8 MDD, and N=6 HC were not able to be analyzed.
  Additionally, N=1 HC was found to have Obstructive sleep apnea, and was thus excluded, and N=1 MDD was found to have had ingested alcohol prior to the experimental night and was thus excluded from analysis.
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Subjects With Major Depressive Disorder | Control
Number analyzed (Participants) | 24 | 13
millivolts (mV)
  MEP at Baseline | 195.07 (99.72) | 179.16 (74.24)
  MEP after slow-wave disruption | 323.22 (286.94) | 212.73 (198.54)
Statistical Analysis 1: Comparison: Subjects With Major Depressive Disorder vs Control; Test type: Other; p < 0.05, ANOVA — a priori threshold for statistical significance set at <0.05; Repeated measures ANOVA, main effect of time, F(1,35) =4.73

2. Primary Outcome: Compare Markers Associated With Plasticity (BDNF) in Individuals With MDD to Healthy Controls
Description: Brain-derived Neurotrophic Factor (BDNF) - Protein found in blood used to measure synaptic plasticity
Time Frame: one month
Population: Due to difficulties with blood collection, data from N=5 MDD, and N=5 HC were not able to be analyzed.
  Additionally, N=1 HC was found to have Obstructive sleep apnea and was thus excluded, and N=1 MDD was found to have had ingested alcohol prior to the experimental night and was thus excluded from analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Subjects With Major Depressive Disorder | Control
Number analyzed (Participants) | 27 | 14
pg/ml
  Plasma BDNF at Baseline | 1599.80 (1010.78) | 1738.32 (1248.35)
  Plasma BDNF after Slow-wave Disruption | 2839.79 (3507.37) | 2860.74 (2590.43)
Statistical Analysis 1: Comparison: Subjects With Major Depressive Disorder vs Control; Test type: Other; p < 0.05, ANOVA — a priori threshold for statistical significance set at p<0.05; Repeated Measures ANOVA, main effect of time, F(1,39) = 4.20

3. Secondary Outcome: Determine if Slow-wave Disruption Alters Mood in Individuals With MDD
Description: Hamilton rating scale for depression - Clinician-administered measure of depression severity.
  The Hamilton Depression Rating Scale is a 17-item, scale that includes questions about depressed mood, suicidal ideation, interest and motivation, irritability, and libido. Participants in this study completed a modified version, the HRSD-NOW (Leibenluft, Moul, Schwartz, Madden, & Wehr, 1993) during the study protocol, which prompts for responses in the context of the present moment and excludes items 4, 5, and 6 (insomnia symptoms), and item 16 (weight loss) which are less appropriate for multi-day assessment. Total scores could range from 0 to 44, with higher scores indicating greater severity of depressive symptomatology.
Time Frame: one month
Population: N=1 HC was found to have Obstructive sleep apnea, and was thus excluded, and N=1 MDD was found to have had ingested alcohol prior to the experimental night and was thus excluded from analysis.
  Additionally, N=1 HC did not complete the HAM-D at one time point and was thus excluded from analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects With Major Depressive Disorder | Control
Number analyzed (Participants) | 32 | 18
score on a scale
  HAM-D at Baseline | 5.25 (2.98) | 1.44 (1.79)
  HAM-D following SWD | 5.53 (3.89) | 1.22 (1.17)
Statistical Analysis 1: Comparison: Subjects With Major Depressive Disorder vs Control; Test type: Other; p < 0.001, ANOVA — a priori threshold for statistical significance set at p <0.05; Repeated measures ANOVA interaction, F(1,48) = 61.849

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Ineligible/Withdrew: Results are reported per Arm/Group, but data from participants who were ineligible or withdrew did not complete the study and therefore had no associated adverse events.
Arm/Group | Control | Subjects With Major Depressive Disorder | Ineligible/Withdrew
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/33 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/33 | 0/11
Other Adverse Events (participants affected / at risk) | 1/20 | 0/33 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=20) | Subjects With Major Depressive Disorder (N=33) | Ineligible/Withdrew (N=11)
Headache (General disorders) | 1 (1) | 0 | 0 — Mild headache

LIMITATIONS AND CAVEATS:
This study was conducted in a sample of individuals with MDD who were relatively young and physically healthy without significant sleep disturbance. Thus, this may not be generalizable to the larger population of individuals with MDD. Cortical excitability was also assessed as a proxy measure of synaptic strength. Because cortical excitability in the MEP of the APB muscle represents more than just synaptic strength, it may not accurately reflect changes in synaptic strength.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT04150718/Prot_SAP_000.pdf